CLINICAL TRIAL: NCT02300896
Title: Functional and Cognitive Impairment Prevention Through Early Physical Activity for Elderly Hospitalized Patients: a Randomized Clinical Trial
Brief Title: Functional and Cognitive Impairment Prevention for Elderly Hospitalized Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23/2014
Record Dates: First submitted 2014-11-19; First posted 2014-11-25 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Functional Impairment; Cognitive Impairment; Elderly
Keywords: exercise; physical fitness; geriatrics
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Group-based exercise training during hospitalization Procedure: Exercise training. Individual program training 5 days a week during hospitalization
  Interventions: Other: Group-based exercise training during hospitalization
- Control (No Intervention): Usual care including rehabilitation when necessary

INTERVENTIONS:
Other: Group-based exercise training during hospitalization — Exercise training. Individual program training 5 days a week during hospitalization
  Arms: Intervention

SUMMARY:
The current model of care for the hospitalized elderly patients has been conditioned by many factors unrelated to the disease process that caused the hospitalization and usually worsen the outcome of hospitalization circumstances. Many times hospitalized elderly patients spend most of the time in bed (even higher than 83% of bed rest versus 4% of those who stand or are walking). These patients have their functional and physiological reserve reduced which makes them more vulnerable to the effects of being bedridden. The consequences are at multiple levels emphasizing the functional loss or cognitive impairment, longer stays, mortality and institutionalization, delirium, deconditioning, pressure ulcers and decreased caloric intake, social isolation, poor quality of life and increased use of resources related to health. Exercise training can prevent functional and cognitive decline and modify even the posterior trajectory.

DETAILED DESCRIPTION:
This study is a randomized clinical trial conducted in a Department of Geriatrics of a tertiary public hospital with 35 beds allocated. Hospitalized patients who meet the inclusion criteria will be randomly assigned to intervention or control group. Patient recruitment will begin in the first 48 hours of admission to the ward, which will be identified through the list of patients admitted to the hospital and assigned to the Department of Geriatrics. The doctor who decides the inclusion in the intervention or control group will not be the attending physician. Patients or their families (if the patient has cognitive impairment) will be informed of the random inclusion in one group, but will not be informed as to which they belong. Randomization will be performed by applying http://www.randomizer.org/. The information in both the intervention group and the control group will obtained in four different stages: the initial visit and at months 3, 6 and 12 after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years and older
* Able to tolerate exercise
* Able to ambulate, with or without personal / technical assistance or move unassisted in a wheelchair
* Able to communicate
* Non-elective admission to hospital

Exclusion Criteria:

* Severe dementia (GDS 7)
* Duration of hospitalization <72 hours
* Unwillingness to either complete the study requirements or to be randomized into control or intervention group
* Unstable cardiovascular disease or other unstable medical condition
* Terminal illness

Min Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Changes in functional status after the intervention (Barthel Index) | Baseline (Hospital Admiission), 1 and 3 months later
  Barthel Index
Changes in functional status after the intervention (Mini Mental State Evaluation, GDS Yesavage, Trail Making Test) | Baseline (Hospital Admiission) and 1 and 3 months later
  Mini Mental State Evaluation, GDS Yesavage, Trail Making Test

SECONDARY OUTCOMES:
Quality of life (EuroQol Scale) | Baseline (Hospital Admission), 1 and 3 months later
  EuroQol Scale
delirium (Confusion Assessment Method, Delirium Rating Scale-Revised-98) | Baseline (Hospital Admission),1 and 3 months later
  Confusion Assessment Method, Delirium Rating Scale-Revised-98
mortality | Baseline (Hospital Admission), 1 and 3 months later
  Days alive since admission to hospital
Use of health resources | Baseline (Hospital Admission), 1 and 3 months later
  New admissions to Hospital, admission to nursing homes, visits to General Practitioner

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Martínez-Velilla, PhD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (1):
- Complejo Hospitalario de Navarra. Department of Geriatrics, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Martinez-Velilla N, Saez de Asteasu ML, Ramirez-Velez R, Zambom-Ferraresi F, Garcia-Hermoso A, Izquierdo M. Recovery of the Decline in Activities of Daily Living After Hospitalization Through an Individualized Exercise Program: Secondary Analysis of a Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2021 Jul 13;76(8):1519-1523. doi: 10.1093/gerona/glab032. PMID 33522565
- [Derived] Ramirez-Velez R, Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Garcia-Hermoso A, Izquierdo M. Handgrip Strength as a Complementary Test for Mobility Limitations Assessment in Acutely Hospitalized Oldest Old. Rejuvenation Res. 2021 Jun;24(3):213-219. doi: 10.1089/rej.2020.2344. Epub 2021 Jan 7. PMID 33267668
- [Derived] Martinez-Velilla N, Valenzuela PL, Saez de Asteasu ML, Zambom-Ferraresi F, Ramirez-Velez R, Garcia-Hermoso A, Librero-Lopez J, Gorricho J, Perez FE, Lucia A, Izquierdo M. Effects of a Tailored Exercise Intervention in Acutely Hospitalized Oldest Old Diabetic Adults: An Ancillary Analysis. J Clin Endocrinol Metab. 2021 Jan 23;106(2):e899-e906. doi: 10.1210/clinem/dgaa809. PMID 33150389
- [Derived] Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Ramirez-Velez R, Garcia-Hermoso A, Izquierdo M. Cognitive Function Improvements Mediate Exercise Intervention Effects on Physical Performance in Acutely Hospitalized Older Adults. J Am Med Dir Assoc. 2021 Apr;22(4):787-791. doi: 10.1016/j.jamda.2020.08.024. Epub 2020 Sep 30. PMID 33011095
- [Derived] Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Ramirez-Velez R, Garcia-Hermoso A, Cadore EL, Casas-Herrero A, Galbete A, Izquierdo M. Changes in muscle power after usual care or early structured exercise intervention in acutely hospitalized older adults. J Cachexia Sarcopenia Muscle. 2020 Aug;11(4):997-1006. doi: 10.1002/jcsm.12564. Epub 2020 Mar 10. PMID 32155323
- [Derived] Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Casas-Herrero A, Cadore EL, Galbete A, Izquierdo M. Assessing the impact of physical exercise on cognitive function in older medical patients during acute hospitalization: Secondary analysis of a randomized trial. PLoS Med. 2019 Jul 5;16(7):e1002852. doi: 10.1371/journal.pmed.1002852. eCollection 2019 Jul. PMID 31276501
- [Derived] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Saez de Asteasu ML, Lucia A, Galbete A, Garcia-Baztan A, Alonso-Renedo J, Gonzalez-Glaria B, Gonzalo-Lazaro M, Apezteguia Iraizoz I, Gutierrez-Valencia M, Rodriguez-Manas L, Izquierdo M. Effect of Exercise Intervention on Functional Decline in Very Elderly Patients During Acute Hospitalization: A Randomized Clinical Trial. JAMA Intern Med. 2019 Jan 1;179(1):28-36. doi: 10.1001/jamainternmed.2018.4869. PMID 30419096
- [Derived] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Suarez N, Alonso-Renedo J, Contin KC, de Asteasu ML, Echeverria NF, Lazaro MG, Izquierdo M. Functional and cognitive impairment prevention through early physical activity for geriatric hospitalized patients: study protocol for a randomized controlled trial. BMC Geriatr. 2015 Sep 15;15:112. doi: 10.1186/s12877-015-0109-x. PMID 26374430